CLINICAL TRIAL: NCT01652508
Title: Individual, Telephone-delivered Acceptance and Commitment Therapy for Smoking Cessation in the Primary Healthcare Setting: Feasibility and Potential Efficacy
Brief Title: Acceptance and Commitment Therapy for Smoking Cessation in the Primary Care Setting
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Yim Wah Mak, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HHSRF9101421
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; Acceptance and Commitment Therapy; primary care setting; randomised controlled trial
MeSH Terms: conditions — Smoking Cessation | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Participants are given printed self-help leaflet on smoking cessation developed by the Department of Health, Hong Kong.
  Interventions: Other: Control
- Acceptance and Commitment Therapy (Experimental): All participants are given a self-help leaflet on smoking cessation. Participants are also given an initial session of face-to-face ACT at a primary health service clinic. In addition, two more subsequent ACT sessions are provided by telephone at one week and one month after the initial intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Other: Control — Participants in the control group are provided a self-help leaflet on smoking cessation only
  Other Names: Control intervention
  Arms: Control
Behavioral: Acceptance and Commitment Therapy — All participants are given an initial smoking cessation session via face to face by Acceptance and Commitment Therapy. Two other sessions using the same therapy will be provided by telephone. The total contact time by ACT will be 45 mins (15 mins per session).
  Arms: Acceptance and Commitment Therapy

SUMMARY:
The purpose of this study is to evaluate the feasibility and potential efficacy of Acceptance and Commitment Therapy (ACT) in enhancing smoking cessation among attendees in primary healthcare settings.

DETAILED DESCRIPTION:
The program is preventive and corrective, and carries brief messages by approaching and influencing services attendees who may not be able to reach in traditional reactive approach method of service users. Those traditional approaches are, for example, quitline and smoking cessation clinic. It can therefore benefit a larger population at low cost.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* currently smoking at least one cigarette per day in the past 30 days
* Hong Kong residents
* able to communicate in Cantonese
* currently residing in Hong Kong and expecting to continue to do so for the next 6 months
* have access to a telephone

Exclusion Criteria:

* currently undergoing another smoking cessation or similar program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence by self report | at 6 months
  self-reports on stopped smoking for a consecutive 7 days proceeding to the assessment at 6 months post-intervention

SECONDARY OUTCOMES:
validated self-report not smoking measured | at 6 months after the baseline
  Obtaining CO measurement and testing urinary cotinine for those participants who report quitting smoking

OTHER OUTCOMES:
Feasibility outcomes | 1 year
  Feasibility outcomes will be assessed in terms of participant recruitment, programme attendance and retention, their acceptance of physical cravings, emotions and thoughts related to smoking

CONTACTS AND LOCATIONS:
Overall Officials: YW Mak, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; AY Loke, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon
  - United Christian Nethersole Community Health Service, Kwong Fuk Community Health Centre, Tai Po, New Territories
  - Heavenly Joy Family Clinic, Tin Shui Wai, New Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mak YW, Lee PH, Loke AY. Predictors of participation in a telephone-based Acceptance and Commitment Therapy for smoking cessation study. BMC Public Health. 2015 Dec 23;15:1288. doi: 10.1186/s12889-015-2650-0. PMID 26701301
- [Result] Mak YW, Loke AY. The acceptance and commitment therapy for smoking cessation in the primary health care setting: a study protocol. BMC Public Health. 2015 Feb 7;15:105. doi: 10.1186/s12889-015-1485-z. PMID 25879419
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Mak YW, Leung DYP, Loke AY. Effectiveness of an individual acceptance and commitment therapy for smoking cessation, delivered face-to-face and by telephone to adults recruited in primary health care settings: a randomized controlled trial. BMC Public Health. 2020 Nov 16;20(1):1719. doi: 10.1186/s12889-020-09820-0. PMID 33198700